CLINICAL TRIAL: NCT05587530
Title: Zero Suicide Implementation and Evaluation in Outpatient Mental Health Clinics
Brief Title: Zero Suicide Implementation in Outpatient Mental Health Clinics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As of 09/2025, the study was unable to be completed due to the administrative pause of research activities at the New York State Psychiatric Institute.
Sponsor: Columbia University (Other)
Collaborators: Research Foundation for Mental Hygiene, Inc. (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lisa Dixon, Edna L. Edison Professor of Psychiatry, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV1378; R56MH112139 (NIH); 8320 (Other: New York State Psychiatric Institute Institutional Review Board); 1383713 (Other: WCG Institutional Review Board)
Record Dates: First submitted 2022-07-29; First posted 2022-10-20 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Suicide
Keywords: Suicide Prevention; Engagement; Retention; Outpatient behavioral health
MeSH Terms: conditions — Suicide; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Informed by data from qualitative participatory interviews and secondary data analysis of administrative databases and based on client and staff stakeholder preferences, the investigators will develop a manualized treatment engagement and retention protocol for suicidal outpatient clients. To determine feasibility and acceptability of the manualized treatment engagement and retention protocol for suicidal outpatient clients, the investigators will conduct a small pilot study with 15 clients across 1-2 clinics (single arm intervention pilot).
Masking Description: N/A - Open pilot trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment engagement and retention intervention for suicidal clients (Experimental): Participants will receive the manualized treatment engagement and retention protocol for suicidal outpatient clients (single-arm intervention pilot). The manualized treatment engagement and retention protocol will be based on client and staff stakeholder preferences, informed by data from qualitative participatory interviews and secondary data analysis of administrative databases (conducted in phase 1).
  Interventions: Behavioral: Treatment engagement and retention intervention for suicidal clients

INTERVENTIONS:
Behavioral: Treatment engagement and retention intervention for suicidal clients — The manualized behavioral intervention for treatment engagement and retention of suicidal clients will be based on client and staff stakeholder preferences, informed by data from qualitative participatory interviews and secondary data analysis of administrative databases (conducted in phase 1). In addition to factors identified by stakeholders, if deemed feasible and acceptable during phase 1, the intervention will include structured phone outreach, shared decision-making, and peer support.

SUMMARY:
The aim of this study is to develop a manualized suicide prevention intervention to improve the retention and engagement of suicidal clients. (For the purposes of this proposal, engagement is defined as return to treatment after the initial session and retention as treatment attendance in an ongoing manner.) In the prior grant received by the investigators (#R01 MH112139) a large-scale project implementing evidence-based suicide prevention practices in 165 outpatient behavioral health clinics in New York State, it was determined that several aspects of the Zero Suicide model were successfully implemented but that treatment engagement and retention of acutely suicidal clients was far from optimal.

This project will have two phases; only the second phase is considered a clinical trial. In the first phase, the investigators will conduct qualitative interviews with clients engaged in outpatient behavioral health for suicide-related reasons, as well as outpatient behavioral health staff (peer specialists and clinicians) with experience working with suicidal clients, to determine to determine client, clinician and situational facilitators and barriers of suicidal clients' engagement in ongoing care. Specifically, interviews will assess if the proposed interventions of shared decision-making (SDM), structured phone outreach (SPO) and peer support are acceptable and feasible from both a client and staff perspective and perceived to be effective in enhancing treatment engagement and retention and decreasing suicidal ideation and behavior. The investigators will also conduct secondary quantitative data analyses with administrative data obtained during the previously-funded project to examine characteristics of those who did not engage or remain in treatment and/or had self-harm behavior during the implementation period, to identify clients who may benefit from additional support or assistance at the outset of treatment and during ongoing care.

In the second phase of the study, the investigators will use the findings from the first phase to develop a manualized treatment engagement and retention protocol and conduct a small pilot study to assess the protocol's feasibility and acceptability to clients and staff (peer specialists and clinicians) and preliminary effectiveness, as indicated by client satisfaction and engagement.

DETAILED DESCRIPTION:
Suicide is the 10th leading cause of death in the US, killing more than 47,000 Americans each year. US suicide deaths have increased dramatically, a staggering 62% increase over the past two decades. While suicide research has made great strides in the development of "best practices" for screening, risk assessment, suicide-specific clinical interventions, and follow-up protocols, there is a striking gap between assessment and intervention development and the implementation of these practices in typical clinical settings.Furthermore, very little research has explored if the "best practices" recommended by clinical experts and researchers are deemed feasible, acceptable, or even desirable by clients experiencing suicidal thoughts and behavior.

ELIGIBILITY:
Inclusion Criteria (clients receiving pilot intervention):

* Age range 18-64 years
* Medicaid eligible
* Currently receiving outpatient behavioral healthcare for suicide-related reasons
* Willingness to participate in the pilot intervention
* Willingness to complete a 1-month follow-up assessment

Inclusion Criteria (peer specialists delivering pilot intervention):

* Any adult participant (18+) is acceptable, though most will be expected to be working age (e.g., 18-65 years old)
* Certified peer specialists working in an outpatient behavioral health setting
* Has experience working with clients enrolled in behavioral healthcare for suicide-related reasons
* Willingness to participate in training and deliver the pilot intervention
* Willingness to complete the pre-training, post-training, and 1-month follow-up assessment

Exclusion criteria (all participants):

* Lacks capacity to consent
* Not fluent to read, write, and/or speak in English

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa B. Dixon, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants progressed beyond Phase 1 (qualitative interviews)
Period: Overall Study
Arm/Group | Treatment Engagement and Retention Intervention for Suicidal Clients
Started | 7
Staff | 5
Clients | 2
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 Staff Participants: Staff members who completed Phase 1 qualitative interviews
- Phase 1 Client Participants: Clients who completed Phase 1 qualitative interviews.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Staff Participants | Phase 1 Client Participants | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Acceptability (Adapted From the Treatment Acceptability and Preference Questionnaire)
Description: Acceptability of the treatment engagement and retention intervention for suicidal clients, as rated by clients receiving the intervention and peer specialists delivering the intervention on an assessment adapted from the Treatment Acceptability and Preference Questionnaire
Time Frame: 1 month
Population: The study was terminated before participants could receive the intervention, therefore no data was collected for this outcome.
Arm/Group | Treatment engagement and retention intervention for suicidal clients
Number analyzed (Participants) | 0

2. Primary Outcome: Feasibility (Adapted From the Treatment Acceptability and Preference Questionnaire)
Description: Feasibility of the treatment engagement and retention intervention for suicidal clients, as rated by clients receiving the intervention and peer specialists delivering the intervention on an assessment adapted from the Treatment Acceptability and Preference Questionnaire
Time Frame: 1 month
Population: as for outcome 1
Arm/Group | Treatment engagement and retention intervention for suicidal clients
Number analyzed (Participants) | 0

3. Primary Outcome: Satisfaction With the Intervention (Adapted From the Treatment Acceptability and Preference Questionnaire)
Description: Satisfaction with the treatment engagement and retention intervention for suicidal clients, as rated by clients receiving the intervention and peer specialists delivering the intervention on an assessment adapted from Treatment Acceptability and Preference Questionnaire
Time Frame: 1 month
Population: as for outcome 1
Arm/Group | Treatment engagement and retention intervention for suicidal clients
Number analyzed (Participants) | 0

4. Secondary Outcome: Perceived Effectiveness
Description: Perceived effectiveness of the treatment engagement and retention intervention for suicidal clients, as rated by clients receiving the intervention and peer specialists delivering the intervention
Time Frame: 1 month
Population: as for outcome 1
Arm/Group | Treatment engagement and retention intervention for suicidal clients
Number analyzed (Participants) | 0

5. Secondary Outcome: Engagement
Description: Rate of return after the first OBH visit for clients assigned to the suicide care pathway, as assessed by Medicaid claims
Time Frame: 1 month
Population: as for outcome 1
Arm/Group | Treatment engagement and retention intervention for suicidal clients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: During qualitative interviews, up to 90 days
Arm/Group | Treatment Engagement and Retention Intervention for Suicidal Clients
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT05587530/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT05587530/ICF_001.pdf